CLINICAL TRIAL: NCT02821026
Title: Allogeneic Islet Cells Transplanted Into the Omentum
Brief Title: Omental Islet Transplant
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00058260
Record Dates: First submitted 2016-06-20; First posted 2016-07-01 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2019-11

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; thymoglobulin; Mycophenolic Acid; Tacrolimus; Etanercept; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Omental islet transplant (Experimental): At the time a suitable islet preparation becomes available, the patient will receive allogeneic islet cells placed in an omental pouch. Islet transplant will be performed under Anti-Thymocyte Globulin induction immunosuppression (5 doses, day -2 prior to transplant to day 2 post-transplant). Maintenance mycophenolate mofetil therapy (1-2 g/day as BID dosing) will be started on Day -1 pre-transplant. Tacrolimus will be administered orally twice daily on Day 1 post-transplant to maintain a trough level of 10-12 ng/mL for 3 months, then 6-10 ng/mL thereafter. Etanercept will be given IV before the islet transplant (50 mg), and then at 25 mg (subcutaneously) on POD +3, +7 and +10. Sirolimus will be used in case of tacrolimus or/and mycophenolate mofetil intolerance.
  Interventions: Procedure: Omental Islet transplant; Drug: Anti-Thymocyte Globulin; Drug: Mycophenolate mofetil; Drug: Tacrolimus; Drug: Etanercept; Drug: Sirolimus

INTERVENTIONS:
Procedure: Omental Islet transplant — The intervention is transplanting the islets into an omental pouch instead of into the liver. The omentum is a large apron-like fold of membrane inside the abdomen that drapes over the intestines. This study will test to see if omental islet transplantation is safe and effective. Standard immunosuppressive medicines (anti-thymocyte globulin, tacrolimus, mycophenolic acid, sirolimus, etanercept) will be used in this study to prevent rejection of the islets.
Drug: Anti-Thymocyte Globulin
  Other Names: Thymoglobulin®
Drug: Mycophenolate mofetil
Drug: Tacrolimus
Drug: Etanercept
Drug: Sirolimus — Sirolimus will be used in case of tacrolimus or/and mycophenolate mofetil intolerance.

SUMMARY:
Islet transplantation is a relatively new procedure used in people with difficult to control Type 1 diabetes. Insulin producing cells (islets) are isolated from a pancreas of a deceased organ donor. After the cells are carefully prepared, the islets are transplanted into patient's body. These transplanted islets may produce insulin for the patient. Patient may be able to reduce or eliminate the need for insulin injections for an unknown period of time. Patients who receive an islet transplant may need to stay on powerful immunosuppressive drugs for as long as the islets remain alive and working. These drugs help to prevent the immune system from attacking the transplanted islets.

Under current standard of care procedure, islets are transplanted into patient's liver. The investigators have learned that some of these cells do not survive the current procedure and are lost around the time of transplant. Therefore in this study, the investigators are studying a new transplant procedure that may help prevent this islet cell loss. The new procedure involves transplanting the islets into an omental pouch instead of into the liver. The omentum is a large apron-like fold of membrane inside the abdomen that drapes over the intestines. This study will test to see if omental islet transplantation is safe and effective. Standard immunosuppressive medicines (anti-thymocyte globulin, tacrolimus, mycophenolic acid, sirolimus, etanercept) will be used in this study to prevent rejection of the islets.

This study is a collaborative research with the University of Miami, and the same study protocol has been in use over there. Recruitment in Edmonton will continue until all subjects [N=6] needed for the study are transplanted. All subjects in this study will receive islet transplants using the study procedure.

DETAILED DESCRIPTION:
BACKGROUND

Current islet transplantation into the portal vein of the liver has shown the unique ability of islets to stabilize blood glucose levels and prevent severe hypoglycemia in a selected group of subjects with type 1 diabetes. The main limitations of islet transplantation are the need for systemic immunosuppression to maintain function and the loss of islet function over time. Additionally, many studies have demonstrated that the current site of transplantation in the liver is not an ideal site due to several factors. These factors include (1) significant liver inflammation following islet infusion; (2) potential for life-threatening procedure-related complications such as bleeding and thrombosis; (3) high levels of immunosuppressive drugs and GI toxins in the liver contributing to islet toxicity; (4) the inability to retrieve islets after infusion; and (5) development of graft dysfunction in a number of recipients of intrahepatic allogeneic and autologous islets.

Based on these premises, development of a clinical protocol for the implantation of islets into the omentum is a desirable goal. As an attempt to maximize the engraftment of islet cell clusters onto the omentum, implantation site should promote islet adherence to the omental peritoneal layer and avoid cell pelleting. Dr. Alejandro's team at University of Miami has recently performed a series of experiments in animal models of diabetes to assess the feasibility of transplanting pancreatic islets in the omentum using a plasma-thrombin gel. With that approach, the islets are re-suspended in either donor or autologous plasma and distributed in the omental pouch (created by sutures) to avoid pelleting. Cell adherence is achieved by addition of clinical-grade recombinant human thrombin that reacts with plasma to create a biocompatible, degradable gel containing the islet graft.

The investigators have outlined the initial patient trial as 6 subjects, based on clinical judgment and extensive experience in clinical islet transplantation trials. If initial safety and efficacy is satisfactory (no adverse events related to the transplantation and efficacy in 2 of the 3 first transplanted subjects), the investigators will transplant 3 additional subjects.

OBJECTIVES

Primary Objective

Safety: To demonstrate the safety of islet transplantation into an omental pouch site for the treatment of subjects with type 1 diabetes (T1D).

Secondary Objective

Efficacy: To demonstrate the efficacy of islet transplantation into an omental pouch site for the treatment of T1D in subjects with hypoglycemia unawareness and a history of severe hypoglycemic episodes.

Primary Endpoints

The primary safety endpoint is to demonstrate patient safety throughout all stages of the trial.

The primary efficacy endpoint is the proportion of subjects with HbA1c ≤6.5% at 1 year AND free of severe hypoglycemic events from Day 28 to Day 365, inclusive, after the islet transplant.

Secondary Endpoints

Secondary efficacy endpoints: At 75±7, 365 ± 14 ,and 730 ± 14 days following the islet transplant(s): the percent reduction in insulin requirements; HbA1c; Mean Amplitude of Glycemic Excursions (MAGE); Lability Index (LI); Ryan hypoglycemia severity (HYPO) score; Clarke score; number of severe hypoglycemic episodes; basal (fasting) and 90-min glucose and c-peptide derived from the mixed-meal tolerance test (MMTT); beta-score; C-peptide creatinine ratio; acute insulin response to glucose (AIRglu), insulin sensitivity, and disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance (FSIGT) test; glucose variability and hypoglycemia duration derived from the continuous glucose monitoring system® (CGMS); and Quality of life (QOL) measures: EuroQol five dimensions questionnaire (EQ-5D), Hypoglycemia Fear Survey (HFS), SF-36v2, Diabetes Distress scale).

Secondary safety endpoints: Safety, including incidence of post-transplant infections, malignancies, morbidity, and other adverse events (AEs) (e.g., increased body weight and hypertension) associated with conventional immunosuppression. Renal function as measured by serum creatinine, glomerular filtration rate (GFR) and other relevant laboratory parameters. Lipid profiles (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol) over time.

At 75 ± 7 and 365 ± 14 days following the islet transplant, and at two years following the final islet transplant: the incidence and severity of AEs related to the islet transplant procedure including: bleeding (>2 g/dL decrease in hemoglobin concentration); wound complication (infection or subsequent hernia); torsion of omentum; gastrointestinal obstruction; abscess; cysts; need for surgical intervention. The incidence and severity of AEs related to the immunosuppression including: allergy; reduction in GFR; addition or intensification of antihyperlipidemic therapy; gastrointestinal toxicity; neutropenia, anemia, or thrombocytopenia; viral, bacterial, or fungal infections; and benign or malignant neoplasms. The incidence of immune sensitization defined by presence of anti-HLA antibodies absent prior to transplantation. The incidence of discontinuation of immunosuppression.

PROCEDURES

Prior to transplantation, the patient is screened, qualified, listed for transplant, and signs the informed consent form.

At the time a suitable islet preparation becomes available, the patient will receive allogeneic islet cells placed in an omental pouch. The details of this surgical procedure will be addressed in Question 5.0.

Islet transplant will be performed under Anti-Thymocyte Globulin (ATG, Thymoglobulin®) induction immunosuppression (5 doses, day -2 prior to transplant to day 2 post-transplant). Maintenance mycophenolate mofetil (MMF) therapy (1-2 g/day as BID dosing) will be started on Day -1 pre-transplant. Tacrolimus will be administered orally twice daily on Day 1 post-transplant to maintain a trough level of 10-12 ng/mL for 3 months, then 6-10 ng/mL thereafter. Etanercept will be given IV before the islet transplant (50 mg), and then at 25 mg (subcutaneously) on post-operative day (POD) +3, +7 and +10.

FOLLOW UP

Subject will undergo a 24-month follow-up period following their islet transplant. 19 study visits during the first year after the transplant, and 4 more study visits during the 2nd year after the transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 to 65 years of age.
2. Ability to provide written informed consent.
3. Mentally stable and able to comply with the procedures of the study protocol.
4. Clinical history compatible with T1D with onset of disease at <40 years of age, insulin-dependence for > 5 years at the time of enrollment, and a sum of subject age and insulin-dependent diabetes duration of ≥28.
5. Absent stimulated c-peptide (<0.3 ng/mL) in response to a MMTT (Boost® 6 mL/kg body weight to a maximum of 360 mL; another product with equivalent caloric and nutrient content may be substituted for Boost®) measured at 60 and 90 min after the start of consumption.
6. Involvement in intensive diabetes management, defined as self-monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist, with at least 3 clinical evaluations during the 12 months prior to study enrollment.
7. At least one episode of severe hypoglycemia in the 12 months prior to study enrollment.
8. Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more OR A HYPO score greater than or equal to the 90th percentile (1047) during the screening period; OR Marked glycemic lability characterized by wide swings in blood glucose (BG) despite optimal diabetes therapy and defined by an LI score greater than or equal to the 90th percentile (43 mmol/L2/h·wk-1) during the screening period; OR A composite of a Clarke score of 3 or less and a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than or equal to the 75th percentile (329) during the screening period.

Exclusion Criteria:

1. Body Mass Index (BMI) >30 kg/m2 or patient weight ≤50 kg.
2. Insulin requirement of >1.0 IU/kg/day or <15 U/day.
3. HbA1c >10%.
4. Untreated proliferative diabetic retinopathy.
5. Blood Pressure: systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg.
6. Measured glomerular filtration rate <80 mL/min/1.73 m2 calculated using the subject's measured serum creatinine and Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation1 or Modification of Diet in Renal Disease [MDRD] study estimation formula). Strict vegetarians (vegans) with a calculated GFR <70 mL/min/1.73m2 are excluded. The absolute (raw) GFR value will be used for subjects with body surface areas >1.73m2
7. Presence or history of macroalbuminuria (>300mg/g creatinine).
8. Presence or history of panel-reactive anti-HLA antibodies above background by flow cytometry.
9. For female subjects: Serum or urine Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. If sexually active, subject must use at least two medically accepted methods of birth control from the following list: oral contraceptives, Norplant®, Depo-Provera®, intrauterine device (IUD), barrier devices with spermicide. Condoms used alone are not acceptable. Instead of the male condom, it is acceptable to use a female condom with one of the other methods for women listed above.
10. Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB) Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
11. Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
12. Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection within one year prior to study enrollment.
13. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
14. Known active alcohol or substance abuse.
15. Baseline Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL). Participants with lymphopenia are allowed if the investigator determines there is no additional risk and obtain clearance from a hematologist.
16. A history of Factor V deficiency.
17. Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an international normalized ratio (INR) >1.5.
18. Severe co-existing cardiac disease, characterized by any one of these conditions:

    1. recent myocardial infarction (within past 6 months).
    2. evidence of ischemia on functional cardiac exam within the last year.
    3. left ventricular ejection fraction <30%.
19. Persistent elevation of liver function tests at the time of study entry. Persistent serum glutamic-oxaloacetic transaminase (SGOT [AST]), serum glutamate pyruvate transaminase (SGPT [ALT]), Alk Phos or total bilirubin, with values >1.5 times normal upper limits will exclude a patient.
20. Symptomatic cholecystolithiasis.
21. Acute or chronic pancreatitis.
22. Symptomatic peptic ulcer disease.
23. Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders potentially interfering with the ability to absorb oral medications.
24. Hyperlipidemia despite medical therapy (fasting low-density lipoprotein [LDL] cholesterol > 130 mg/dL (3.36 mmol/L), treated or untreated; and/or fasting triglycerides > 200 mg/dL (2.26 mmol/L)).
25. Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
26. Treatment with any anti-diabetic medications other than insulin within 4 weeks of enrollment.
27. Use of any investigational agents within 4 weeks of enrollment.
28. Administration of live attenuated vaccine(s) within 2 months of enrollment.
29. Any medical condition that, in the opinion of the investigator, will interfere with the safe participation in the trial.
30. Treatment with any immunosuppressive regimen at the time of enrollment.
31. A previous islet transplant.
32. A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and the transplant occurred more than 6 months prior to enrollment.
33. Inflammatory bowel disease.
34. History of intestinal obstructions.
35. Previous major abdominal surgery.
36. History of peritonitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
The incidence of Serious Adverse Events | 2 years following islet transplant
The proportion of subjects with HbA1c ≤ 6.5% at 1 year AND free of severe hypoglycemic events from Day 28 to Day 365, inclusive, after the islet transplant | From Day 28 to Day 365 inclusive after islet transplant

SECONDARY OUTCOMES:
The percent reduction in insulin requirements at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
The percent reduction in insulin requirements at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
The percent reduction in insulin requirements at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in HbA1c at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in HbA1c at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in HbA1c at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in Mean Amplitude of Glycemic Excursions at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in Mean Amplitude of Glycemic Excursions at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in Mean Amplitude of Glycemic Excursions at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in Lability Index at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in Lability Index at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in Lability Index at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in Ryan hypoglycemia severity score at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in Ryan hypoglycemia severity score at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in Ryan hypoglycemia severity score at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in Clarke score at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in Clarke score at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in Clarke score at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in number of severe hypoglycemic episodes at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in number of severe hypoglycemic episodes at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in number of severe hypoglycemic episodes at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in basal (fasting) and 90- min glucose and c-peptide derived from the mixed-meal tolerance test at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in basal (fasting) and 90- min glucose and c-peptide derived from the mixed-meal tolerance test at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in basal (fasting) and 90- min glucose and c-peptide derived from the mixed-meal tolerance test at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in beta-score at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in beta-score at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in beta-score at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in C-peptide creatinine ratio at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in C-peptide creatinine ratio at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in C-peptide creatinine ratio at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in acute insulin response to glucose at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in acute insulin response to glucose at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in acute insulin response to glucose at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in insulin sensitivity at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in insulin sensitivity at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in insulin sensitivity at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance (FSIGT) test at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance (FSIGT) test at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in disposition index derived from the insulin-modified frequently-sampled intravenous glucose tolerance (FSIGT) test at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in glucose variability and hypoglycemia duration derived from the continuous glucose monitoring system® (CGMS) at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in glucose variability and hypoglycemia duration derived from the continuous glucose monitoring system® (CGMS) at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in glucose variability and hypoglycemia duration derived from the continuous glucose monitoring system® (CGMS) at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in diabetes distress scores measured by Diabetes Distress scale at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in diabetes distress scores measured by Diabetes Distress scale at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in diabetes distress scores measured by Diabetes Distress scale at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in health status measured by EQ-5D at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in health status measured by EQ-5D at Day 365± 14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in health status measured by EQ-5D at Day 730± 14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in the score measured by Hypoglycemia Fear Survey-HFS at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in the score measured by Hypoglycemia Fear Survey-HFS at Day 365±14after islet transplant | Baseline and Day 365± 4 after islet transplant
Change from baseline in the score measured by Hypoglycemia Fear Survey-HFS at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Change from baseline in health scores obtained through SF-36v2 health survey at Day 75±7 after islet transplant | Baseline and Day 75±7 after islet transplant
Change from baseline in health scores obtained through SF-36v2 health survey at Day 365±14 after islet transplant | Baseline and Day 365±14 after islet transplant
Change from baseline in health scores obtained through SF-36v2 health survey at Day 730±14 after islet transplant | Baseline and Day 730±14 after islet transplant
Incidence of AEs associated with conventional immunosuppression | 2 years following islet transplant
Renal function (serum creatinine and GFR) | Day 75 ± 7, Day 365 ± 14 and Day 730± 14 after islet transplant
Lipid profiles (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol) | Day 75 ± 7, Day 365 ± 14 and Day 730± 14 after islet transplant
The incidence of AEs related to the islet transplant procedure | 2 years following islet transplant
The incidence of immune sensitization defined by presence of anti-HLA antibodies absent prior to transplantation | 2 years following islet transplant
The incidence of discontinuation of immunosuppression | 2 years following islet transplant

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, Principal Investigator — University of Alberta
Locations (1):
- Clinical Islet Transplant Program, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Islet Transplant Program — http://www.islet.ca